CLINICAL TRIAL: NCT01751919
Title: A Randomized, Open-label, Single-dose, Crossover Clinical Trial to Compare the Pharmacokinetics of Imatinib Mesylate Tablet 400 mg (1 Tablet) and Glivec Film-coated Tablet 100 mg (4 Tablets) After Oral Administration in Healthy Male Subjects (Phase I)
Brief Title: A Clinical Trial to Compare the Pharmacokinetics of Imatinib Mesylate Tablet 400mg (1 Tablet) and Glivec Film-coated Tablet 100mg (4 Tablets)(Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Imatinib_CML_I
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Myeloid Leukemia; Gastrointestinal Stromal Tumor
Keywords: CML; GIST
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (RT) (Other): * Period 1: Glivec film-coated tablet 100 mg, 4 tablets (Active comparator)
  * Period 2: Imatinib mesylate tablet 400 mg, 1 tablet (experimental)
  Interventions: Drug: Imatinib mesylate tablet 400 mg, 1 Tablet; Drug: Glivec film-coated tablet 100 mg, 4 Tablets
- Group 2 (TR) (Other): * Period 1: Imatinib mesylate tablet 400 mg, 1 tablet (experimental)
  * Period 2: Glivec film-coated tablet 100 mg, 4 tablets (Active comparator)
  Interventions: Drug: Imatinib mesylate tablet 400 mg, 1 Tablet; Drug: Glivec film-coated tablet 100 mg, 4 Tablets

INTERVENTIONS:
Drug: Imatinib mesylate tablet 400 mg, 1 Tablet
Drug: Glivec film-coated tablet 100 mg, 4 Tablets

SUMMARY:
1. Investigational Product

   1. Imatinib mesylate tablet 400 mg
   2. Glivec film-coated tablet 100 mg (Comparator)
2. Expected target disease

   1. chronic myeloid leukemia
   2. Gastrointestinal stromal tumors
3. Study design : Randomized, open-label, single dose, two-period, two-way, crossover study

   1. 36 healthy subjects, 2 groups (18 subjects/group)
   2. 2 Period (either 1-a(1 tablet) or 1-b(4 tablet))
   3. wash-out period : 14 days
4. Evaluation on pharmacokinetics(PKs) and safety

   1. PKs : Cmax, AUClast, Tmax, AUCinf, t1/2
   2. safety : adverse events, physical examination, vital sign, ECG, Laboratory test
5. Statistical method

   1. Demography Characteristics
   2. Pharmacokinetic parameters
   3. Safety data

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers between the ages of 20 to 50 years old
* weight more than 55kg and within the range of ±20% of ideal body weight (IBW)
* having neither congenital/chronic diseases nor pathological symptoms/findings as results of medical examination
* doctor determines to be suitable as subjects within 3 weeks ago before administration

Exclusion Criteria:

* Hypersensitivity(or history of hypersensitivity) to medicines including imatinib mesylate
* Active Liver Diseases or exceed 1.5 times the normal range of AST, ALT, total bilirubin
* Creatinine clearance < 80 mL/min
* Gastrointestinal diseases or surgeries that affect absorption of drug
* Excessive drinking(exceed 21units/week)
* Smoking over 10 cigarettes per day

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum concentration in plasma (Cmax) of Imatinib mesylate | Pre-dose(0h) AND 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 h post-dose
Area under the plasma concentration-time curve from zero time until the last measurable concentration (AUClast) of Imatinib mesylate | Pre-dose(0h) AND 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 h post-dose

SECONDARY OUTCOMES:
Time to Cmax (Tmax) of Imatinib mesylate | Pre-dose(0h) AND 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 h post-dose
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) of Imatinib mesylate | Pre-dose(0h) AND 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 h post-dose
Terminal Elimination Half-life (t1/2) of Imatinib mesylate | Pre-dose(0h) AND 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University, Daegu, South Korea

REFERENCES:
- [Background] Parrillo-Campiglia S, Ercoli MC, Umpierrez O, Rodriguez P, Marquez S, Guarneri C, Estevez-Parrillo FT, Laurenz M, Estevez-Carrizo FE. Bioequivalence of two film-coated tablets of imatinib mesylate 400 mg: a randomized, open-label, single-dose, fasting, two-period, two-sequence crossover comparison in healthy male South American volunteers. Clin Ther. 2009 Oct;31(10):2224-32. doi: 10.1016/j.clinthera.2009.10.009. PMID 19922893
- [Background] Nikolova Z, Peng B, Hubert M, Sieberling M, Keller U, Ho YY, Schran H, Capdeville R. Bioequivalence, safety, and tolerability of imatinib tablets compared with capsules. Cancer Chemother Pharmacol. 2004 May;53(5):433-8. doi: 10.1007/s00280-003-0756-z. PMID 15132131